CLINICAL TRIAL: NCT01163604
Title: Phase 4 Study of Argatroban for Preventing Occlusion and Restenosis After Intracranial and Extracranial Artery Stenting
Brief Title: Argatroban for Preventing Occlusion and Restenosis After Intracranial and Extracranial Artery Stenting
Acronym: APORIAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Xinfeng Liu, Jinling Hospital, China, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JLH
Record Dates: First submitted 2010-06-28; First posted 2010-07-16 (Estimated); Results first posted 2014-11-07 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-10

CONDITIONS: CVD
Keywords: Argatroban; intracranial artery stenting; extracranial artery stenting; occlusion; restenosis
MeSH Terms: conditions — Bites and Stings | interventions — argatroban; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Argatroban group (Experimental): Patients who underwent intracranial and extracranial artery stenting were randomly chosen to receive continuous infusions of argatroban for 2 days before and 3 days after stenting, with accompanied aspirin and clopidogrel treatment.
  Interventions: Drug: Argatroban
- non-argatroban treated group (Experimental): Patients who underwent intracranial and extracranial artery stenting were randomly chosen to receive only aspirin and clopidogrel treatment.
  Interventions: Drug: non-argatroban treated group

INTERVENTIONS:
Drug: Argatroban — Intravenous Infusion, 20mg/day for 2 days before and 3 days after stenting, (10mg/3h, twice a day), with accompanied aspirin and clopidogrel treatment
  Other Names: Argartroban
  Arms: Argatroban group
Drug: non-argatroban treated group — Patients who underwent intracranial and extracranial artery stenting were randomly chosen to receive only aspirin and clopidogrel treatment.
  Other Names: aspirin, clopidogrel
  Arms: non-argatroban treated group

SUMMARY:
Argatroban is a selective thrombin inhibitor, and previous study had suggested that argatroban use post PCI could potentially prevent reocclusion. But there has no study on large sample of argatroban treated restenosis post cranial stenting. This study will test the safety and efficacy of the argatroban on prevent occlusion and restenosis in patients with intracranial and extracranial artery stenting.

DETAILED DESCRIPTION:
The risk of restenosis post intracranial and extracranial artery stenting is 20-40%, therefore, in the past, aspirin and clopidogrel were performed as anticoagulant therapy post stenting.But this treatment had limited effectiveness upon restenosis. Argatroban is a selective thrombin inhibitor, and previous study had suggested that argatroban use post PCI could potentially prevent reocclusion. But there has no study on large sample of argatroban treated restenosis post cranial stenting. This study will test the safety and efficacy of the argatroban on prevent occlusion and restenosis in patients with intracranial and extracranial artery stenting.

ELIGIBILITY:
Inclusion Criteria:

* For extracranial artery lesion, stenting was considered for symptomatic stenosis≥50% or asymptomatic stenosis≥70%; according to intracranial artery lesion, stenting was considered for symptomatic stenosis≥70% in invalid patients after intensive medical therapy.
* Successfully had intracranial or extracranial artery stenting

Exclusion Criteria:

* Evidence of hemorrhagic brain infarction, intracranial and extracranial hematoma, or intraventricular hemorrhage, or Gastrointestinal ulcers in 3 months
* Hypersensitivity to contrast agent
* Malignant hypertension
* Difficult to perform the intracranial and extracranial artery stenting
* Severe hepatic or cardiac disorders, infectious disorders, dehydration, etc.
* Serum creatinine >1.5 mg/dL
* Hypersensitivity to test drugs
* Difficult to hand follow-up visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xinfeng Liu, MD, Study Chair — Department of Neurology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Department of Neurology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The present study was a single-center, open-label, prospective, randomized, controlled pilot one. Enrollment of participants began in August 2010, and completed in August 2011. The local ethics committee approved the study, and written informed consent was obtained in all recruited patients.
Pre-assignment Details: The present study was a single-center, open-label, prospective, randomized, controlled pilot one. Enrollment of participants began in August 2010, and completed in August 2011. The local ethics committee approved the study, and written informed consent was obtained in all recruited patients.
Groups:
- "Aspirin" and "Clopidogrel" Interventions Group: Patients who underwent intracranial and extracranial artery stenting were randomly chosen to receive only aspirin and clopidogrel treatment.
  non-argatroban treated group: Patients who underwent intracranial and extracranial artery stenting were randomly chosen to receive only aspirin and clopidogrel treatment.
Period: Overall Study
Arm/Group | Argatroban Group | "Aspirin" and "Clopidogrel" Interventions Group
Started | 58 (August 2010) | 56 (August 2010)
Completed | 58 (August 2011) | 56 (August 2011)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Argatroban Group | Non-argatroban Treated Group | Total
Number analyzed (Participants) | 58 | 56 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.07 (11.87) | 28.14 (11.46) | 28.10 (11.64)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 56 | 114
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 51 | 51 | 102
Region of Enrollment [Number; unit: participants]
  China | 58 | 56 | 114

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Occlusion and Restenosis at One Year
Description: Stenosis detected by DSA(digital subtraction angiography),CTA(CT angiography)or MRA(MR angiography)was measured according to NASCET(North American Symptomatic Carotid Endarterectomy Trial)method.Concretely, NASCET stenosis is calculated from the ratio of the linear luminal diameter of the narrowest segment of the diseased portion of the artery to the diameter of the artery beyond any poststenotic dilatation: NASCET=(1-md/C)×100%
Time Frame: at one year
Measure: Number; unit: participants
Arm/Group | Argatroban Group | Non-argatroban Treated Group
Number analyzed (Participants) | 58 | 56
participants | 58 | 56

2. Secondary Outcome: NIHSS, mRS
Description: NIHSS and mRS are widely used stroke deficit assessment tools. Most clinical stroke-related trials require a baseline and outcome severity assessment. The baseline of mRS is rank 0, NIHSS 0; the severity of mRS is 6, NIHSS 42. AS many patients have one or more strokes before they perform stenting, this study selected NIHSS and mRS as the supplementary materials to estimate the stroke deficit of patients and to reflect the therapeutic effect and safety of stenting and argatroban therapy. These two scales are performed according to the guidance before and after stenting and argatroban therapy.
Time Frame: at one year
Reporting Status: Not Posted

3. Secondary Outcome: Various Adverse Effects
Time Frame: at one year
Reporting Status: Not Posted

4. Secondary Outcome: Clinical Endpoints
Time Frame: at one year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1year
Description: Serious and Other [Non-Serious] Adverse Events were not collected
Arm/Group | Argatroban Group | Non-argatroban Treated Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes